CLINICAL TRIAL: NCT00856622
Title: A 6-Month, Randomized, Double-Masked Comparison Of Fixed Combination Of Latanoprost And Timolol With The Individual Components, Continuing Into A 6-Month Open Label Safety Study Of Fixed Combination In Patients With Glaucoma Or Ocular Hypertension.
Brief Title: A Study Demonstrating The Effect Of Latanoprost In Combination With Timolol, Latanoprost Alone And Timolol Alone On Eye Pressure In Open Angle Glaucoma Or Ocular Hypertension In Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96TIPG004; A6641005
Record Dates: First submitted 2009-03-02; First posted 2009-03-06 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2018-10

CONDITIONS: Ocular Hypertension; Glaucoma; Open-angle Glaucoma
Keywords: open-angle glaucoma ocular hypertension glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma; Glaucoma, Open-Angle | interventions — Xalacom; Timolol; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed combination of latanoprost 0.005% and timolol 0.5% (Experimental)
  Interventions: Drug: i. Fixed combination of latanoprost 0.005% and timolol 0.5%
- timolol 0.5% ophthalmic solution (Active Comparator): one drop in the morning and evening
  Interventions: Drug: timolol 0.5% ophthalmic solution
- latanoprost 0.005% ophthalmic solution (Active Comparator): placebo in the morning and latanoprost .005% in the evening
  Interventions: Drug: latanoprost 0.005% ophthalmic solution

INTERVENTIONS:
Drug: i. Fixed combination of latanoprost 0.005% and timolol 0.5% — one drop in the morning and placebo in the evening
  Other Names: xalacom, xalcom
  Arms: Fixed combination of latanoprost 0.005% and timolol 0.5%
Drug: timolol 0.5% ophthalmic solution — one drop in the morning and evening
  Other Names: timoptic
  Arms: timolol 0.5% ophthalmic solution
Drug: latanoprost 0.005% ophthalmic solution — placebo in the morning and latanoprost .005% in the evening
  Other Names: xalatan
  Arms: latanoprost 0.005% ophthalmic solution

SUMMARY:
The purpose of this study is to demonstrate that fixed combination of latanoprost and timolol (PhXA41) has better IOP lowering effect than the individual monotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary open angle glaucoma, capsular glaucoma, pigmentary glaucoma or ocular hypertension.
* Patients currently on IOP reducing therapy: IOP greater than or equal to 25mmHg (two IOP determinations at pre-study separated by at least one hour) OR Patients without IOP reducing therapy: IOP greater than or equal to 30mmHg (two IOP determinations at pre-study separated by at least one hour).

Exclusion Criteria:

* History of acute angle closure or closed/barely open anterior chamber angle.
* Current use of contact lenses.
* Ocular surgery or argon laser trabeculoplasty (ALT) within three months prior to pre-study visit.
* Ocular inflammation/infection occurring within three months prior to pre-study visit.
* Hypersensitivity to benzalkonium chloride or to any other component of the study drug solutions.
* Other abnormal ocular condition or symptom preventing the patient from entering the study, according to the investigator's judgement.
* Cardiac failure, sinus bradycardia, second and third degree of atrioventricular block. (The routines for prescribing topical B-blocking agents will be followed.
* Bronchial asthma, history of bronchial asthma or chronic obstructive pulmonary disease. (The routines for prescribing topical B-blocking agents will be followed).
* Pregnancy
* Women of childbearing potential who has not used adequate contraceptive methods during the last three months.
* Inability to adhere to treatment/visit plan.
* Have participated in any other clinical study within one month prior to pre-study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 1997-08; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate that the fixed combination of latanoprost and timolol has a better IOP-reducing effect than the individual monotherapies. | 6 months

SECONDARY OUTCOMES:
To examine, within treatment groups, the diurnal IOP reducing effect from baseline for all treatments at Week 26 | 6 Months
To compare the diurnal IOP reducing effect from baseline between the monotherapies latanoprost and timolol at Week 26 | 6 Months
To compare the number of treatment failures and patients withdrawn due to uncontrolled IOP from baseline to Week 26 between treatment groups | 6 Months
To compare the proportion of patients reaching pre-specified (15, 18, and 21 mmHg) target diurnal IOPs between the treatment groups at Week 26 | 6 Months
To describe the IOP development from baseline to Week 26 for all treatment groups | 6 Months
To compared the IOP reducing effect from baseline to Week 26 of the monotherapies with the IOP reducing effect from Week 26 to Week 52 of the fixed combination | 6 Months
To examine, within the fixed combination treatment group, the diurnal IOP reducing effect from baseline to Week 26 and Week 52 | 6 Months
To follow the safety variables throughout the study periods. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- Germany (34):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Aalen
  - Pfizer Investigational Site, Ahaus
  - Pfizer Investigational Site, Alzey
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Abbach
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Coesfeld
  - Pfizer Investigational Site, Dillingen
  - Pfizer Investigational Site, Eitorf
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Freising
  - Pfizer Investigational Site, Fulda
  - Pfizer Investigational Site, Greifswald
  - Pfizer Investigational Site, Gummersbach
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Hirschaid
  - Pfizer Investigational Site, Iserlohn
  - Pfizer Investigational Site, Koblenz
  - Pfizer Investigational Site, Leonberg
  - Pfizer Investigational Site, Leverkusen
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Mülheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Offenbach
  - Pfizer Investigational Site, Osnabrück
  - Pfizer Investigational Site, Parsberg
  - Pfizer Investigational Site, Siegburg
  - Pfizer Investigational Site, Sulzbach
  - Pfizer Investigational Site, Trier
  - Pfizer Investigational Site, Weiden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=96TIPG004